CLINICAL TRIAL: NCT03688646
Title: Randomised Control Trial Study To Compare The Efficacy of ONS Supplementation With Standard Dietary Advice On Nutritional Outcome in HNC Outpatients Undergoing Treatment in Radiotherapy Clinic
Brief Title: Efficacy of ONS Supplementation in HNC Outpatient Under Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Malaysia (Other Government)
Responsible Party: Principal Investigator, Norshariza Jamhuri, Clinical Dietitian, Principal Investigator, National Cancer Institute, Malaysia
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: NMRR-15-2171-28670
Record Dates: First submitted 2018-08-31; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intensive nutrition intervention group receiving standardised oral nutrition supplement provided once daily throughout cancer treatment with 4 session of dietary consultation by designated dietitian for monitoring of diet intake and diet modification to meet patient's requirement
  Interventions: Dietary Supplement: Intensive Nutrition Intervention
- Control group (No Intervention): Routine care were given to this group inclusive of 4 session of dietary consultation by designated dietitian for monitoring of diet intake and diet modification to meet patient's requirement and also prescription of oral nutrition supplement where needed. Oral nutrition supplement was not provided

INTERVENTIONS:
Dietary Supplement: Intensive Nutrition Intervention
  Arms: Intervention group

SUMMARY:
A RCT study to compare the efficacy of ONS supplementation with standard dietary advice on nutritional outcome inHNC outpatients undergoing treatment in radiotherapy clinic. IThe study population are all adult HNC outpatients receiving radiotherapy with or without chemotherapy treatments at Radiotherapy Clinic,NCI. Selected patient will be randomized into Control Group and Intervention Group until each group have 20 subjects, where the total of sample will be 40 patients (in consideration of 50% dropouts) and data will be collected at baseline (prior to treatment), week 2, 4, and the final data will be at week 6 or final day of cancer treatment. Study objectives are to determine the efficacy of ONS supplementation in outpatient HNC undergoing treatment in Radiotherapy Clinic, NCI, to determine nutritional outcome (weight loss and BMI, body composition, dietary intake, albumin and hemoglobin level), functional outcome (handgrip strength) and side effect outcome (nutrition impact symptoms) in HNC outpatients given intensive nutrition intervention with outpatients given routine care. This study also want to find association of Intensive nutrition intervention versus routine care in nutrition outcome, functional and side effect outcome in both group. Subjects in intervention group will received standardize ONS supplementation every day during treatments once daily with frequent dietary advice accordingly to the patients condition while control group will received standard routine care which includes frequent dietary advice without supplementation of ONS. Study hypothesis is there is no significant difference in nutritional outcome, functional outcome and side effect outcome between HNC outpatients receiving INI when compared to HNC outpatient receiving routine care undergoing radiotherapy treatment. There is also no association between these two groups in nutritional outcome, functional outcome and side effect outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Those who diagnosed with Head and Neck Cancer (HNC) and receiving radiotherapy with or without chemotherapy treatments.
2. Able to communicate.
3. Patient admitted to ward less than 5 days.

Exclusion Criteria:

1. Patient on tube feeding.
2. Patient was already on ONS before study period.
3. Patient already started treatments (referring to chemotherapy, radiotherapy and CCRT) before study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
nutritional outcome (weight changes) | 7 weeks
  changes of outcome within and between group weight in kilogram measurement are taken during baseline, 2nd weeks, 4th weeks and 6th weeks of treatment
functional outcome | 7 weeks
  preliminary handgrip strength and changes handgrip strength in kilogram force instrument: handgrip dynamometer measurement taken during baseline, 2nd week, 4th weeks and 6th weeks of treatment instrument: body composition analyzer changes of outcome within and between group
side effect outcome | 7 weeks
  changes of nutrition impact symptoms experienced by patients within and between group instrument: validated HSNC© checklist measured during baseline, 2nd weeks, 4th weeks, and 6th weeks of treatment
nutritional outcome (body composition) | 7 weeks
  muscle mass in kilogram body fat mass in kilogram measurement taken during baseline, 2nd week, 4th weeks and 6th weeks of treatment instrument: body composition analyzer changes of outcome within and between group
nutritional outcome (biochemical data - albumin and hemoglobin level) | 7 weeks
  albumin in g/L hemoglobin in g/dL measurement taken during baseline, 2nd week, 4th weeks and 6th weeks of treatment instrument: body composition analyzer changes of outcome within and between group
nutritional outcome (body mass index) | 7 weeks
  body mass in kilogram/meter2 measurement taken during baseline, 2nd week, 4th weeks and 6th weeks of treatment instrument: body composition analyzer changes of outcome within and between group

CONTACTS AND LOCATIONS:
Overall Officials: Norshariza Jamhuri, Principal Investigator — National Cancer Institute (NCI)

IPD SHARING:
Plan to Share IPD: No